CLINICAL TRIAL: NCT02325544
Title: COgnitive Behavioural Therapy Versus Standardised Medical Care for Adults With Dissociative Non-Epileptic Seizures: A Multicentre Randomised Controlled Trial (CODES)
Brief Title: Comparing Different Treatments in Reducing Dissociative Seizure Occurrence
Acronym: CODES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: University of Edinburgh (Other); University of Sheffield (Other); University of Sussex (Other); South London and Maudsley NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CSP 136836
Record Dates: First submitted 2014-12-15; First posted 2014-12-25 (Estimated); Last update posted 2020-10-09 (Actual); Status verified 2016-02

CONDITIONS: Convulsion, Nonepileptic; Conversion Disorder; Dissociative Disorder
Keywords: dissociative seizures,; psychogenic nonepileptic seizures
MeSH Terms: conditions — Seizures; Conversion Disorder; Dissociative Disorders; Psychogenic Nonepileptic Seizures | interventions — Cognitive Behavioral Therapy; Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CBT+SMC (Experimental): 12 sessions of Cognitive Behavioural Therapy adapted for DS (plus one booster session) plus standardised medical care
  Interventions: Behavioral: Cognitive Behavioral Therapy; Behavioral: Standardized Medical Care
- SMC (Active Comparator): Standardised medical care provide by neurologist and/or psychiatrist
  Interventions: Behavioral: Standardized Medical Care

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — 12 sessions of CBT (over 4-5 months) +1 booster session. Guided by a therapy manual and patient handouts; will involve setting homework tasks. Although treatment is manualised, it allows treatment to be formulation-based i.e. tailored to the person.
  Standardised medical as described in other intervention.
  Arms: CBT+SMC
Behavioral: Standardized Medical Care — Delivered by neurologists/ psychiatrists - both will be involved in discussing diagnosis. It will Include an information sheet about dissociative seizures and direction to self-help websites, general information provision about management of DS and support, consideration of psychiatric comorbidities / associated drug treatment and general review but no CBT techniques.
  Other Names: Treatment as usual

SUMMARY:
The study will test the hypothesis that Cognitive Behavioural Therapy plus Standardised Medical Care (SMC) will have greater clinical and cost effectiveness than SMC alone in treating adult patients with dissociative seizures which had not initially ceased after diagnosis.

About 12-20% of patients who attend neurology or specialist epilepsy clinics because of seizures do not in fact have epilepsy. Most of these people have what are referred to as dissociative (non-epileptic) seizures (DS). This means that they have episodes that resemble epileptic seizures but which have no medical reason for their occurrence and instead are due to psychological factors. In younger adults DS are about four times more common in women than men. A high percentage of these people will have other psychological or psychiatric problems and may have other medically unexplained symptoms. It is generally thought that people with DS will benefit from psychological treatments. However, studies on this have been small or have not compared the psychological therapy with the treatment people normally receive (standardised medical care). There is some evidence that cognitive behavioural therapy (CBT), which is a widely accepted talking therapy that focuses on the person's thoughts, emotions and behaviour, as well as considering the physical reactions and sensations that may occur in people's bodies, may lead to a reduction in how often people have DS. The investigators have previously developed a CBT package for people with DS. In a relatively small study by our group, published in 2010, people receiving CBT overall showed greater reduction in how often they had their DS. The investigators are now conducting a larger study, across several different hospitals, to obtain more definite results about the effectiveness of our CBT approach for DS.

The investigators aim to invite ~ 500 adult patients with DS (but without current active epilepsy), who have been given their diagnosis by a neurologist or specialist in epilepsy, to take part in their study. Up to 698 might be invited if insufficient patients are progressing to the RCT.

The investigators will collect initial information about these people and ask them to keep a record of how often they have their DS following diagnosis. Three months after the diagnosis, those who have agreed to take part in the study will be seen by a psychiatrist, who will undertake a psychiatric assessment and ask them about factors which may have led to the development of their DS. Patients who have continued to have DS in the previous 8 weeks and who meet other eligibility criteria and are willing to take part in the trial, will be randomly allocated to standardised medical care or CBT (plus standardised medical care) as further treatment for their seizures. These people will be asked to continue to complete seizure diaries and questionnaires, provide regular seizure frequency data following receipt of DS diagnosis and will need to be willing to attend weekly/fortnightly sessions if allocated to CBT. The investigators initially aim to randomise 298 people (149 to each study arm) although now allow for up to 356 to account for loss to follow-up.

DETAILED DESCRIPTION:
There is an initial observational phase to this study followed by a parallel group, two-arm multi-centre pragmatic randomised controlled trial (interventional phase).

In the observational phase patients will be given their diagnosis of dissociative seizures by a neurologist/epilepsy specialist and will be told about the CODES study. In addition to a leaflet on dissociative seizures they will, if interested in the study and are willing to be referred to a psychiatrist, be given an information sheet about DS and about the study and the doctor will document their agreement to be contacted by a research nurse/worker. This person will arrange to contact them, clarify study details, obtain informed consent, collect demographic details and explain seizure diary recording. They will then contact the patient fortnightly (bi-weekly)for seizure data. The investigators initially aim to recruit ~500 patients at this stage.

After 3 months the patient will be reviewed by a neuropsychiatrist/ liaison psychiatrist/ psychiatrist with interest in DS who will undertake a clinical assessment, review the patient's eligibility for the interventional phase of the study and if eligible will explain the RCT. Patients will be given a further leaflet on DS and a Participant Information Sheet and the psychiatrist will document interested patients' willingness to again be contacted by a research nurse/worker. That person will then explain the RCT in greater detail, obtain informed consent, undertake a baseline assessment including a MINI and instruct patients to keep seizure records for which data will be collected fortnightly. .Randomisation of between 298 and 356 people (depending on follow-up rates) to either CBT plus standardised medical care (SMC) or to SMC alone will occur after informed consent has been obtained and baseline measures have been collected. The stratification factor will be liaison/neuropsychiatry centre. The research workers and trial statistician will remain blinded. Computer-generated randomisation will be conducted remotely (for more details see www.ctu.co.uk - randomisation - advanced) by the King's Clinical Trials Unit (KCTU) at the Institute of Psychiatry, Psychology and Neuroscience. The investigators will maintain strict allocation concealment. The investigators will test the RWs' blinding by asking them to record when they think that allocation was revealed and record the group to which they thought patients had been allocated.

CBT will be delivered over 12 sessions (each approximately one hour in length) over a 4-5 month period with one booster session at 9 months post randomisation. The investigators' treatment model has been developed from a single case study, trialled in an open label study and then in a Pilot RCT. The model is based on the two-process fear escape-avoidance model and conceptualises DS as dissociative responses to cues (cognitive/emotional/physiological or environmental) that may (but not in all cases) have been associated with profoundly distressing or life-threatening experiences, such as abuse or trauma, at an earlier stage in the person's life and which have previously produced intolerable feelings of fear and distress. Written handouts supplement the content of face-to face therapy sessions. The investigators will record therapy sessions and undertake treatment fidelity ratings. Therapists will receive training prior to treating study patients.

Neurologists and psychiatrists with an interest in DS will deliver standardised medical care (SMC). They will have guidelines as to the delivery of standardised medical care. Information leaflets will be given to the patients. The research team will provide this material. SMC by psychiatrists will include support, consideration of psychiatric comorbidities and any associated drug treatment and general review but no CBT techniques.

The investigators allow for some local variation in the number of neurology and psychiatry SMC sessions after randomisation.

Measures will be recorded at baseline, six months and 12 months post randomisation. In addition to quantitative analyses, a nested qualitative study will investigate experiences of CBT and SMC and factors acting as facilitators and barriers to participation, as well as of healthcare professionals'.experiences of delivering the study.

ELIGIBILITY:
Inclusion Criteria:

1. The inclusion criteria applied at the initial recruitment stage will be as follows:

   * adults (≥18yrs) with DS that have continued to occur within the previous 8 weeks and have been confirmed by video EEG telemetry or, where not achievable, clinical consensus; patients who have chronic DS can be included if they have been seen by the relevant Study Neurologist who has reviewed their diagnosis and communicated this to them according to the Study protocol
   * ability to complete seizure diaries and questionnaires;
   * willingness to complete seizure diaries regularly and undergo psychiatric assessment 3 months after DS diagnosis;
   * no documented history of intellectual disabilities;
   * ability to give written informed consent.
2. Inclusion criteria evaluated at the randomisation stage will be as follows:

   * adults (≥18yrs) with DS initially recruited at point of diagnosis;
   * willingness to continue to complete seizure diaries and questionnaires;
   * provision of regular seizure frequency data following receipt of DS diagnosis;
   * willingness to attend weekly/fortnightly sessions if randomised to CBT
   * both clinician and patient think that randomisation is acceptable
   * ability to give written informed consent.

Exclusion Criteria:

The exclusion criteria applied at the initial recruitment stage will be as follows:

* having a diagnosis of current epileptic seizures as well as DS. Patients with both DS and ES have been included in small studies but there is no method for verifying that patients can accurately differentiate between epileptic seizures and DS;
* inability to keep seizure records or complete questionnaires independently;
* meeting DSM-IV criteria for current drug/alcohol dependence;
* insufficient command of English to later undergo CBT without an interpreter or to complete questionnaires independently. Reasons for this include the need to self-rate secondary outcomes using scales not validated for non-English speaking populations, the considerable cost and uncertainty of being able reliably to engage sufficiently competent interpreters, and the need to demonstrate the delivery of therapy in terms of quality and manual adherence.
* having previously undergone a CBT-based treatment for dissociative seizures at a trial participating centre
* currently having CBT for another disorder, if this will not have ended by the time that the psychiatric assessment takes place.

Exclusion criteria evaluated at the randomisation stage will be as follows:

* current epileptic seizures as well as DS, for reasons given above;
* not having had any DS in the 8 weeks prior to the psychiatric assessment, 3 months post diagnosis;
* having previously undergone a CBT-based treatment for dissociative seizures at a trial participating centre
* currently having CBT for another disorder
* active psychosis;
* meeting DSM-IV criteria for current drug/alcohol dependence; this may exacerbate symptoms/alter psychiatric state and health service use and affect recording of seizures;
* current benzodiazepine use exceeding the equivalent of 10mg diazepam/day;
* the patient is thought to be at imminent risk of self harm, after (neuro)psychiatric assessment or structured psychiatric assessment by the Research Worker with the MINI, followed by consultation with the psychiatrist.
* known diagnosis of Factitious Disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 368 (Actual)
Dates: Start 2014-10-01; Primary Completion 2017-05-31 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Change in seizure frequency | Outcome assessed at 12 month post randomisation,
  Monthly DS frequency

SECONDARY OUTCOMES:
Change in informant rating | Outcome assessed at 12 month post randomisation only
  A rating by an informant as to whether compared to study entry seizure frequency is worse the same better or whether they are seizure free; data collected 6 & 12 months post randomisation; 6 month measures are only collected for data modelling and to maintain participant involvement but the trial endpoint was measured at 12 months only;
Change in self-rated seizure severity | Outcome assessed at 12 month post randomisation only
  Two items from the Seizure Severity Scale (Cramer et al., 2002), asking how severe and bothersome DS were in the past month; data collected at baseline (recorded pre-randomisation) , 6 & 12 months post randomisation; 6 month measures are only collected for data modelling and to maintain patient involvement but the trial endpoint was measured at 12 months only.
Seizure freedom | Outcome assessed at 12 month post randomisation only
  Patient's self-reported longest period of seizure freedom between the 6- and 12-month follow-up and whether or not the patient is seizure free in the last 3 months of the trial; data collected 12 months post randomisation; the trial endpoint was measured at 12 months only.
>50% reduction in seizure frequency | Outcome assessed at 12 month post randomisation only
  The number of patients in each group who at the 6- and 12-month follow-up show >50% reduction in seizure frequency, compared to baseline (pre-randomisation); data collected at baseline and 6 & 12 months post randomisation; 6 month measures are only collected for data modelling and to maintain patient involvement but the trial endpoint was measured at 12 months only.
Change in Quality of life (QoL) | Outcome assessed at 12 month post randomisation only
  Health-related QoL using the SF-12v2 (Ware et al.,1996); data collected at baseline (recorded pre-randomisation) , 6 & 12 months post randomisation; 6 month measures are only collected for data modelling and to maintain patient involvement but the trial endpoint was measured at 12 months only.
Change in QALYs | Outcome assessed at 12 month post randomisation only
  We will use EQ-5D-5L (EuroQol group, 1990), a 5-domain, 5-level, multi-attribute scale collected at baseline (recorded pre-randomisation) , 6 & 12 months post randomisation; 6 month measures are only collected for data modelling and to maintain patient involvement but the trial endpoint was measured at 12 months only.
Change in psychosocial functioning | Outcome assessed at 12 month post randomisation only
  Work and Social Adjustment Scale (Mundt et al 2002) collected at baseline (recorded pre-randomisation) , 6 & 12 months post randomisation; 6 month measures are only collected for data modelling and to maintain patient involvement but the trial endpoint was measured at 12 months only.
Change in psychiatric symptoms and psychological distress | Outcome assessed at 12 month post randomisation only
  We will measure anxiety, depression and somatisation with the GAD7 (Spitzer et al., 2006), PHQ9 (Kroenke et al., 2001) and an extended PHQ15 (Kroenke et al., 2002; Sharpe et al., 2010), derived from the Patient Health Questionnaire which reflects DSM-IV diagnoses. We will also use a general measure of psychological distress, the CORE-10 (Connell & Barkham, 2007); this assesses self-reported global psychological distress; data collected at baseline (recorded pre-randomisation) , 6 & 12 months post randomisation; 6 month measures are only collected for data modelling and to maintain patient involvement but the trial endpoint was measured at 12 months only.
Change in patients self-rated global outcome and satisfaction with treatment | Outcome assessed at 12 month post randomisation only
  CGI Clinical Global Impression (Guy 1976) change score yields a self-rated global measure collected at 6 & 12 months post randomisation; 6 month measures are only collected for data modelling and to maintain patient involvement but the trial endpoint was measured at 12 months only.
Clinician rating of change | Outcome assessed at 12 month post randomisation only
  The CGI change scale will be rated by CBT therapists at the end of session 12 and by the SMC doctor at the 12-month follow-up.
Change in health service use and informal care (self-report) | Outcome assessed at 12 month post randomisation only
  Adapted Client Service Receipt Inventory (Beecham & Knapp, 2001); data collected at baseline (recorded pre-randomisation) , 6 & 12 months post randomisation; 6 month measures are collected for data modelling and to give a total health service use over the 12 months of the post-randomisation period and to maintain patient involvement but the trial endpoint was measured at 12 months only.
Change in health service use | Outcome assessed at 12 months post randomisation
  Linkage data sets from NHS Health and Social Care Information Centre (Hospital Episode Statistics) eDRIS (NHS National Services Scotland Information Services Division (ISD) and Wales (NHS Wales Informatics Service)

CONTACTS AND LOCATIONS:
Overall Officials: Laura H Goldstein, PhD MPhil, Principal Investigator — King's College London
Locations (40):
- United Kingdom (40):
  - Derbyshire Community Health Services Nhs Trust, Bakewell
  - Birmingham and Solihull Mental Health Nhs Foundation Trust, Birmingham
  - University Hospital Birmingham Nhs Foundation Trust, Birmingham
  - Berkshire Healthcare Nhs Foundation Trust, Bracknell
  - Brighton and Sussex University Hospitals Nhs Trust, Brighton
  - Cambridge University Hospitals Nhs Foundation Trust, Cambridge
  - Cambridgeshire and Peterborough Nhs Foundation Trust, Cambridge
  - East Kent Hospitals University Nhs Foundation Trust, Canterbury
  - Cardiff and Vale University Local Health Board, Cardiff
  - Chesterfield Royal Hospital Nhs Foundation Trust, Chesterfield
  - Dartford and Gravesham Nhs Trust, Dartford
  - Derbyshire Healthcare Nhs Foundation Trust, Derby
  - NHS Lothian, Edinburgh
  - Medway Nhs Foundation Trust, Gillingham
  - Leeds Partnerships Nhs Foundation Trust, Leeds
  - Leeds Teaching Hospitals Nhs Trust, Leeds
  - Barts and the London Nhs Trust, London
  - East London Nhs Foundation Trust, London
  - University College London Hospitals Nhs Foundation Trust, London
  - Royal Free Hampstead Nhs Trust, London
  - Guy'S and St Thomas' Nhs Foundation Trust, London
  - Lewisham Healthcare Nhs Trust, London
  - South London and Maudsley NHS Foundation Trust, London
  - King'S College Hospital Nhs Foundation Trust, London
  - St George'S Healthcare Nhs Trust, London
  - South West London and St George'S Mental Health Nhs Trust, London
  - Imperial College Healthcare Nhs Trust, London
  - Maidstone and Tunbridge Wells Nhs Trust, Maidstone
  - The Newcastle Upon Tyne Hospitals NHS Trust, Newcastle
  - Northumberland Tyne and Wear NHS Foundation Trust, Newcastle upon Tyne
  - Royal Berkshire Nhs Foundation Trust, Reading
  - East Sussex Healthcare Nhs Trust, Saint Leonards-on-Sea
  - Sheffield Health and Social Care Nhs Foundation Trust, Sheffield
  - Sheffield Teaching Hospitals Nhs Foundation Trust, Sheffield
  - University Hospital Southhampton NHS Trust, Southampton
  - Croydon Health Services Nhs Trust, Thornton Heath
  - West London Mental Health Nhs Foundation Trust, Uxbridge
  - Kent and Medway Nhs and Social Care Partnership Trust, West Malling
  - Western Sussex Hospitals Nhs Trust, Worthing
  - Sussex Partnership Nhs Foundation Trust, Worthing

REFERENCES:
- [Background] Goldstein LH, Chalder T, Chigwedere C, Khondoker MR, Moriarty J, Toone BK, Mellers JD. Cognitive-behavioral therapy for psychogenic nonepileptic seizures: a pilot RCT. Neurology. 2010 Jun 15;74(24):1986-94. doi: 10.1212/WNL.0b013e3181e39658. PMID 20548043
- [Background] Goldstein LH, Mellers JD, Landau S, Stone J, Carson A, Medford N, Reuber M, Richardson M, McCrone P, Murray J, Chalder T. COgnitive behavioural therapy vs standardised medical care for adults with Dissociative non-Epileptic Seizures (CODES): a multicentre randomised controlled trial protocol. BMC Neurol. 2015 Jun 27;15:98. doi: 10.1186/s12883-015-0350-0. PMID 26111700
- [Background] Robinson EJ, Goldstein LH, McCrone P, Perdue I, Chalder T, Mellers JDC, Richardson MP, Murray J, Reuber M, Medford N, Stone J, Carson A, Landau S. COgnitive behavioural therapy versus standardised medical care for adults with Dissociative non-Epileptic Seizures (CODES): statistical and economic analysis plan for a randomised controlled trial. Trials. 2017 Jun 6;18(1):258. doi: 10.1186/s13063-017-2006-4. PMID 28587649
- [Background] Jordan H, Feehan S, Perdue I, Murray J, Goldstein LH. Exploring psychiatrists' perspectives of working with patients with dissociative seizures in the UK healthcare system as part of the CODES trial: a qualitative study. BMJ Open. 2019 May 9;9(5):e026493. doi: 10.1136/bmjopen-2018-026493. PMID 31072856
- [Background] Goldstein LH, Robinson EJ, Reuber M, Chalder T, Callaghan H, Eastwood C, Landau S, McCrone P, Medford N, Mellers JDC, Moore M, Mosweu I, Murray J, Perdue I, Pilecka I, Richardson MP, Carson A, Stone J; CODES Study Group. Characteristics of 698 patients with dissociative seizures: A UK multicenter study. Epilepsia. 2019 Nov;60(11):2182-2193. doi: 10.1111/epi.16350. Epub 2019 Oct 13. PMID 31608436
- [Background] Goldstein LH, Robinson EJ, Mellers JDC, Stone J, Carson A, Chalder T, Reuber M, Eastwood C, Landau S, McCrone P, Moore M, Mosweu I, Murray J, Perdue I, Pilecka I, Richardson MP, Medford N; CODES Study Group. Psychological and demographic characteristics of 368 patients with dissociative seizures: data from the CODES cohort. Psychol Med. 2021 Oct;51(14):2433-2445. doi: 10.1017/S0033291720001051. Epub 2020 May 11. PMID 32389147
- [Background] Wilkinson M, Day E, Purnell J, Pilecka I, Perdue I, Murray J, Hunter EM, Goldstein LH. The experiences of therapists providing cognitive behavioral therapy (CBT) for dissociative seizures in the CODES randomized controlled trial: A qualitative study. Epilepsy Behav. 2020 Apr;105:106943. doi: 10.1016/j.yebeh.2020.106943. Epub 2020 Feb 18. PMID 32078929
- [Background] Read J, Jordan H, Perdue I, Purnell J, Murray J, Chalder T, Reuber M, Stone J, Goldstein LH. The experience of trial participation, treatment approaches and perceptions of change among participants with dissociative seizures within the CODES randomized controlled trial: A qualitative study. Epilepsy Behav. 2020 Oct;111:107230. doi: 10.1016/j.yebeh.2020.107230. Epub 2020 Jul 5. PMID 32640411
- [Background] Stone J, Callaghan H, Robinson EJ, Carson A, Reuber M, Chalder T, Perdue I, Goldstein LH. Predicting first attendance at psychiatry appointments in patients with dissociative seizures. Seizure. 2020 Jan;74:93-98. doi: 10.1016/j.seizure.2019.11.014. Epub 2019 Nov 28. PMID 31869756
- [Result] Goldstein LH, Robinson EJ, Mellers JDC, Stone J, Carson A, Reuber M, Medford N, McCrone P, Murray J, Richardson MP, Pilecka I, Eastwood C, Moore M, Mosweu I, Perdue I, Landau S, Chalder T; CODES study group. Cognitive behavioural therapy for adults with dissociative seizures (CODES): a pragmatic, multicentre, randomised controlled trial. Lancet Psychiatry. 2020 Jun;7(6):491-505. doi: 10.1016/S2215-0366(20)30128-0. Epub 2020 May 20. PMID 32445688
- [Derived] Goldstein LH, Robinson EJ, Chalder T, Stone J, Reuber M, Medford N, Carson A, Moore M, Landau S. Moderators of cognitive behavioural therapy treatment effects and predictors of outcome in the CODES randomised controlled trial for adults with dissociative seizures. J Psychosom Res. 2022 Jul;158:110921. doi: 10.1016/j.jpsychores.2022.110921. Epub 2022 Apr 19. PMID 35617911
- [Derived] Goldstein LH, Robinson EJ, Pilecka I, Perdue I, Mosweu I, Read J, Jordan H, Wilkinson M, Rawlings G, Feehan SJ, Callaghan H, Day E, Purnell J, Baldellou Lopez M, Brockington A, Burness C, Poole NA, Eastwood C, Moore M, Mellers JD, Stone J, Carson A, Medford N, Reuber M, McCrone P, Murray J, Richardson MP, Landau S, Chalder T. Cognitive-behavioural therapy compared with standardised medical care for adults with dissociative non-epileptic seizures: the CODES RCT. Health Technol Assess. 2021 Jun;25(43):1-144. doi: 10.3310/hta25430. PMID 34196269
- See also: CODES study website — http://www.codestrial.org/